CLINICAL TRIAL: NCT07128290
Title: PErioperative CISGEM + Rilvegostomig in High-Risk Resectable Intra Hepatic CholangioCarcinoma Phase II Single Arm Study - Multicenter
Brief Title: PErioperative CISGEM + Rilvegostomig in High-Risk Resectable Intra Hepatic CholangioCarcinoma
Acronym: PEHRICCA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 118 - FFCD 2402; 2025-521302-17-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-13; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc)
Keywords: Perioperative; Rilvegostomig; CISGEM; High-risk resectable; intrahepatic cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CISGEM + Rilvegostomig (Experimental): RILVEGOSTOMIG : For each cycle one administration at D1 every 3 weeks 750 mg IV administration over 60 minutes (up to a total of 90 minutes).
  CISGEM: For each cycle administration at D1 and D8 every 3 weeks
  * Cisplatine 25 mg/m² in 1 hour IV in 1000 ml NaCl 0,9 % then 500 ml NaCl 0,9 %
  * Gemcitabine 1000 mg/m² en 30 mn IV dans 250 ml NaCl 0,9 %
  Interventions: Drug: CISGEM + Rilvegostomig

INTERVENTIONS:
Drug: CISGEM + Rilvegostomig — Administration of 4 cycles pre-operative and 4 cycles post-operative of Cisplatine associated to Gemcitabine with rilvegostomig
  RILVEGOSTOMIG : For each cycle one administration at D1 every 3 weeks
  • 750 mg IV administration over 60 minutes (up to a total of 90 minutes). CISGEM: For each cycle administration at D1 and D8 every 3 weeks
  * Cisplatine 25 mg/m² in 1 hour IV in 1000 ml NaCl 0,9 % then 500 ml NaCl 0,9 %
  * Gemcitabine 1000 mg/m² en 30 mn IV dans 250 ml NaCl 0,9 %

SUMMARY:
The goal of this trial is to determine whether the combination of CISGEM and Rilvegostomig during the perioperative period works to improve outcomes of patient undergoing surgery of high-risk of intrahepatic cholangiocarcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. WHO Performance Status 0-1
3. Body weight > 30kg
4. Histo/cytologically proven intrahepatic cholangiocarcinoma.
5. Measurable disease as defined by RECIST 1.1 criteria (Response Evaluation Criteria in Solid Tumors).
6. Naive to systemic treatment and loco regional treatment for biliary tract cancer
7. At least one of the following high-risk criteria of post resection relapse:

   * Tumor Size ≥ 50 mm and/or multiple nodules
   * cN+
   * Risk of narrow margin (< 10 mm)
   * Macrovascular invasion
8. Adequate organ function, as defined by the following:

   * Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) ≤ 2,5 x Upper Limit of Normal (ULN)
   * Total serum bilirubin ≤ 1.5 ULN This will not apply to patients with confirmed Gilbert's syndrome
   * Prothrombin ratio > 70 % and/or Factor V > 70 % in case of oral anticoagulation therapy
   * Serum albumin ≥ 30 g/L
   * Haemoglobin ≥ 10 g/dl and no transfusion within 4 weeks before inclusion
   * Absolute Neutrophil Count (ANC) ≥ 1.5 G/L
   * Platelets ≥ 150 G/L
9. Creatinine clearance ≥ 45 ml/min (calculated by CKD - EPI formula)
10. Life expectancy ≥ 3 months
11. Female postmenopausal for at least one year or surgically infertile for at least 6 weeks, or highly effective contraception for male and female patients of childbearing potential for the duration of study and for 7 months after the last dose of drug for female and 4 months for male.
12. A negative pregnancy test for inclusion for all female patients of child-bearing potential.
13. Patient covered by a plan of the French Social Security system.
14. Written informed consent obtained from the patient prior to performing any protocol-related procedures
15. Patient with available tumor tissue sample for the study or willing to have a biopsy

Exclusion Criteria:

1. Existence of metastases or distant lymph node involvement considered as metastatic
2. Locally advanced disease considered as definitively non resectable
3. Cirrhosis with Child Pugh ≥ B7

   1. Any history of liver decompensation: hepatic encephalopathy, presence of ascites
   2. Presence of clinically significant portal hypertension (platelets counts < 150G/L and/or liver stiffness > 20kPa and/or presence of oesophageal and/or gastric varices)
4. Mixed histology (hepatocholangiocarcinoma)
5. Persistent toxicities (> grade 2 NCI-CTCAE version 5.0) caused by previous cancer therapy.
6. Contraindication to immunotherapy: Active or prior documented autoimmune or inflammatory disorders or any severe or uncontrolled systemic disease
7. Current or prior use of immunosuppressive medication within 14 days before the first dose of protocol treatment
8. History of allogenic organ transplantation
9. Known or suspected allergy or hypersensitivity to any of the study drugs or any of the study drug excipients (cisplatin, gemcitabine and Rilvegostomig)
10. Live vaccine administration within 30 days prior to the first dose of study treatment Note: Patients, if enrolled, should not receive live vaccine whilst receiving investigational product and up to 6 months after the last dose of investigational product.
11. Uncontrolled infection with human immunodeficiency virus (HIV). Required conditions for inclusion are as follows: undetectable viral RNA, CD4+ count ≥350 cells/μL no history of AIDS-defining opportunistic infection within the past 12 months, stable condition for at least 4 weeks on the same anti-HIV medications.
12. Active and untreated infection with hepatitis B and/or hepatitis C Note: Patients with past HBV infection or resolved HBV infection (defined as having a negative HBsAg test and a positive hepatitis B core antigen [HBc] antibody test) are eligible.
13. Other active cancer or history of cancer within 2 years, except for carcinoma in situ of the cervix or basal cell or squamous cell skin carcinoma or any other carcinoma in situ, considered cured
14. History of clinically significant arrhythmia, cardiomyopathy of any etiology; symptomatic congestive heart failure (as defined by New York Heart Association class ≥ 3), history of myocardial infarction within the past 6 months. Participation in another clinical study with an investigational product during the last 4 weeks
15. Pregnant or breastfeeding woman.
16. Person deprived of liberty or under guardianship or incapable of giving consent
17. Inability to undergo the medical follow-up of the trial for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients alive without progression at 12 months | 12 months after inclusion
  Progression was assessed by the investigator according to RECIST
  1.1 criteria based on imaging studies performed every 9 weeks, Clinical progressions, not confirmed on imaging, were not be counted in the primary endpoint.
  Death for all causes is also an event.

SECONDARY OUTCOMES:
Overall survival | Up to 24 months after inclusion
  Overall survival is defined as the time from the date of inclusion to the patient's death (all causes). For alive patients, the date of the last news will be taken into account.

CONTACTS AND LOCATIONS:
Overall Officials: Gael ROTH, Dr, Principal Investigator — CHU DE GRENOBLES ALPES
Locations (9):
- France (9):
  - Chu Caen Normandie, Caen
  - Centre Gf Leclerc, Dijon
  - Chu de Dijon, Dijon
  - Chu Grenoble Alpes, Grenoble
  - Chu Dupuytren, Limoges
  - Hopital de La Timone Ap-Hm, Marseille
  - Nancy Chru, Nancy
  - Hopital Prive Du Confluent, Nantes
  - Chu de Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: Undecided